CLINICAL TRIAL: NCT04001491
Title: Evaluation of the Interest of 18F-FDG Positron Emission Tomography in the Management of Unexplained Fevers and Inflammatory Syndromes in Elderly Subjects
Brief Title: Interest of 18F-FDG Positron Emission Tomography in the Management of Fevers and Inflammatory Syndromes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7473
Record Dates: First submitted 2019-06-25; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Inflammation
Keywords: Inflammation; Inflammatory syndromes; fever; Tomography; Positron emission at 18F-FDG; Elderly patients; Internal medicine; Pet-Scan
MeSH Terms: conditions — Inflammation; Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients aged 75 and over represent a heterogeneous population with fragile subjects who have a higher risk of poor tolerance to many tests and especially who have a risk of major functional loss in the event of hospitalization. It is therefore necessary to adapt our prescriptions and not to impose on these patients an examination that is unnecessary. Or on the contrary, not to do without, out of ignorance, a minimally invasive examination that could be useful to these patients.

In this study, the investigators wish to evaluate the interest of the Pet-Scan in the therapeutic management of these elderly patients

ELIGIBILITY:
Inclusion criteria:

* Patient aged 75 years and over,
* Patients cared for at the HUS, in hospital or in consultation, during the defined period (from 01/05/2013 to 31/12/2018)
* Having had an 18FDG-PET/TDM
* For fever or inflammatory syndrome check-ups, regardless of the duration of the evolution and the examinations already carried out
* Patient who has not expressed opposition to the reuse of their data for the purposes of this research.

Exclusion criteria:

* Patient who has expressed opposition to participating in the study
* Known explanation for fever or inflammatory syndrome
* Subjects under legal protection
* Subject under the protection of justice
* Subject under guardianship or curatorship

Translated with www.DeepL.com/Translator

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient treated at the University Hospitals of Strasbourg for a check-up of fever or inflammatory syndrome, regardless of the duration of the evolution and the examinations already carried out
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the interest of the Pet-Scan in the therapeutic management of subjects aged 75 years and over with unexplained fever or inflammatory syndrome. | 1 month
  That is, to assess whether or not the therapeutic course of action has been modified by this examination, resulting in either the discontinuation or initiation of medical, surgical or radiotherapy treatment

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel ANDRES, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de Médecine Interne, diabète et maladies métaboliques - Médicale B, Strasbourg, France